CLINICAL TRIAL: NCT02522897
Title: Evaluation of the "Treat-and-extend" Scheme in Patients With Retinal Vein Occlusion (RVO) With and Without LASER Treatment of Ischaemic Retinal Areas
Acronym: PEARL
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: PD. Dr. med. Armin Wolf (Other)
Collaborators: University Hospital, Bonn (Other)
Responsible Party: Sponsor-Investigator, PD. Dr. med. Armin Wolf, PD Dr. med. Armin Wolf, Ludwig-Maximilians - University of Munich
Organization: Ludwig-Maximilians - University of Munich (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EXT-201302-Pearl
Record Dates: First submitted 2015-08-04; First posted 2015-08-13 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Central Retinal Vein Occlusion With Macular Edema
MeSH Terms: interventions — Ranibizumab; Lasers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ranibizumab (Active Comparator): Patients receive intravitreal injections of 0,5 mg Ranibizumab (Lucentis®) / injection following the "treat-and-extend" scheme for 12 months.
  Interventions: Drug: Ranibizumab
- Ranibizumab + Laser (Experimental): Apart from receiving intravitreal injections of 0,5 mg Ranibizumab (Lucentis®) / injection following the "treat-and-extend" scheme for 12 months, patients receive a panretinal photocoagulation on visit 3 and / or 4.
  Interventions: Drug: Ranibizumab; Device: Laser

INTERVENTIONS:
Drug: Ranibizumab
  Other Names: Lucentis
Device: Laser
  Other Names: Visulas 532s Laser
  Arms: Ranibizumab + Laser

SUMMARY:
The purpose of this study is to determine if additional panretinal photocoagulation of ischemic areas following retinal vein occlusion (RVO) may reduce the rate of recurrence and allow longer treatment intervals in anti-Vascular Endothelial Growth Factor (VEGF) treatment following the "trea-and-extend" scheme.

DETAILED DESCRIPTION:
Patients with macular edema following RVO receive an anti-VEGF treatment by injection of Ranibizumab for 12 months in the "treat-and-extend" scheme. Following this scheme, all patients receive a series of three injections at the interval of 4 weeks. Thereafter, the retreatment interval is determined by results of certain examinations.

The next control including a reinjection is scheduled with an extension of one week until the patient presents signs of recurrence. Assuming that by the time of recurrence the interval is too long, the next control (following a retreatment) is then scheduled one week sooner than the last control. Following this treatment schedule, the individualized retreatment interval is thereafter kept steady.

Half the patients receive an additional panretinal photocoagulation on visit 3 and / or 4. Aim of this study is to investigate if this additional panretinal photocoagulation may result in a longer individualized retreatment interval corresponding to a reduced rate of recurrence of macular edema.

ELIGIBILITY:
Inclusion Criteria:

* retinal vein occlusion with OCT-diagnosed macular edema with a documented duration of 3 months or less
* age over 18
* documented maximal visual acuity of 0,5 ETDRS
* voluntary participation in this study as proven by written informed consent
* ability to follow study instructions and likely to attend and complete all required visits
* pre-menopausal female patients with childbearing potential must use an approved contraceptive method (Pearl index <1)
* pre-menopausal female patients with childbearing potential: a negative serum pregnancy test must be obtained prior to treatment start
* ischemic area of more than 5 pupillary distance (PD) in angiography

Exclusion Criteria:

* subject without legal capacity who is unable to understand the nature, scope, significance and consequences of this clinical trial
* patients with known allergy to Ranibizumab or ingredients of the injection solution
* treatment in another clinical trial with therapeutic intervention or use of any other investigational medicinal product (IMP) during the trial or within the 30 days before enrolment
* known or persistent abuse of medication, drugs or alcohol
* women who are pregnant or breast-feeding
* failure of laboratory inclusion criteria
* diabetic retinopathy
* previous anti-VEGF (Lucentis ®, Avastin®, Eylea®) or LASER therapy due to RVO
* previous intravitreal steroid therapy
* status post excision of the vitreous body
* status post intraocular surgery within 3 months before enrolment
* established or suspected ocular or periocular infection
* evidence of giant cell arteriitis
* retinal hemorrhages that seem to prevent a Laser-treatment of ischemic areals within the following 12 weeks
* unregulated hypertension above 200/120 mmHg
* cerebral vascular occurence or myocardium infarct within 12 months before enrolment
* relevant systemic diseases that might be associated with elevated VEGF serum concentration
* active malignancies (status post successful treatment of malignancies is no exclusion criterion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-08; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Differences in the length of the treatment-free interval in patients with or without panretinal photocoagulation | within 12 months after first injection of Ranibizumab
  Length of the longest interval between reinjections that did not result in recurrence

SECONDARY OUTCOMES:
Number of Injections | within 12 months after first injection of Ranibizumab
Retinal thickness in µm measured by spectral domain (SD)-Optical coherence tomography (OCT) at end-of-study visit | 4-9 weeks after last injection within
  end-of-study visit is performed at individualized retreatment interval (can range from 4-9 weeks) after last injection within 12 months after first injection of Ranibizumab
Visus at end-of-study visit | 4-9 weeks after last injection within
  end-of-study visit is performed at individualized retreatment interval (can range from 4-9 weeks) after last injection within 12 months after first injection of Ranibizumab
Percentage of patients with retinal thickness of more than 220 µm in the OCT examination at the end-of-study visit | 4-9 weeks after last injection within
  end-of-study visit is performed at individualized retreatment interval (can range from 4-9 weeks) after last injection within 12 months after first injection of Ranibizumab

CONTACTS AND LOCATIONS:
Overall Officials: Armin Wolf, PD Dr., Principal Investigator — Eye Clinic of the Ludwig Maximilians University of Munich